CLINICAL TRIAL: NCT00193349
Title: Phase II Evaluation of Gleevec Combined With Camptosar Plus Paraplatin in Patients With Previously Untreated Extensive Stage SCLC
Brief Title: Gleevec Combined With Camptosar Plus Paraplatin in Previously Untreated Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry); Pharmacia and Upjohn (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 59; CSTI571BUS66; CPTAIV-0020-403
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2008-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Imatinib Mesylate; Irinotecan; Carboplatin

INTERVENTIONS:
Drug: Imatinib
Drug: Irinotecan
Drug: Carboplatin

SUMMARY:
This study will evaluate combination chemotherapy for patients with extensive stage small cell lung cancer combined with the potentially useful growth inhibiting effects of Gleevec.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

* Irinotecan + Carboplatin + Imatinib

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Small cell lung cancer with extensive stage disease confirmed by biopsy
* Measurable or evaluable disease
* Ability to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney
* No active brain metastasis.
* No previous chemotherapy or radiation therapy
* Give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Limited stage disease (includes IA, IB, IIA, IIB, and IIIA)
* Active brain metastasis
* Age < 18 years old
* History of a prior malignancy within three years
* Women pregnant or lactating.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate
Response duration

SECONDARY OUTCOMES:
Time to progression
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Simons L, Meng C, Burris HA 3rd, Yardley DA, Grapski R, Schreeder M, Mallidi PV, Greco FA; Minnie Pearl Cancer Research Network. Irinotecan, carboplatin, and imatinib in untreated extensive-stage small-cell lung cancer: a phase II trial of the Minnie Pearl Cancer Research Network. J Thorac Oncol. 2007 Sep;2(9):854-61. doi: 10.1097/JTO.0b013e31814617b7. PMID 17805064
- See also: Published article in the Journal of Thoracic Oncology — http://journals.lww.com/jto/pages/articleviewer.aspx?year=2007&issue=09000&article=00013&type=abstract